CLINICAL TRIAL: NCT04280185
Title: Multicenter Prospective Randomized Controlled Clinical Trial of Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Stage IIc-IV Epithelial Ovarian Cancer After Primary Cytoreductive Surgery
Brief Title: HIPEC in the Treatment of Stage IIc-IV Epithelial Ovarian Cancer After CRS (HIPECOC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cxj2019001434
Record Dates: First submitted 2019-10-15; First posted 2020-02-21 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2019-10

CONDITIONS: Ovarian Cancer; Hyperthermic Intraperitoneal Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperthermic Intraperitoneal chemotherapy (Experimental): Hyperthermic Intraperitoneal chemotherapy was started immediately after CRS, or the first HIPEC was completed within 48 hours after surgery: temperature 43℃, duration 60 minutes, Paclitaxel (60mg/m2) was selected. The second HIEPC was completed 7 days after the first HIPEC: temperature 43℃, duration 60min, carboplatin AUC (5-6) was selected. 30 minutes before using Paclitaxel, 10ML saline + 10mg dexamethasone intravenous infusion, 20mg diphenhyramine intramuscular injection, and 100ML saline + 0.3g cimetidine intravenous infusion. On the eighth day, intravenous chemotherapy with Paclitaxel (135mg/m2) was finally completed. 5 courses of TC intravenous chemotherapy were performed after 3 weeks
  Interventions: Procedure: Hyperthermic Intraperitoneal Chemotherapy
- intravenous chemotherapy (No Intervention): intravenous chemotherapy were performed 6 Cycles after CRS. Paclitaxel: 175mg/m2, iv infusion, no less than 3h per infusion, followed by carboplatin: AUC 5-6, iv infusion, no less than 1h per infusion, 1 dose on the first day of a week, 1 cycle every 3 weeks, a total of 6 cycles. Paclitaxel should be pretreated to prevent severe allergic reactions.

INTERVENTIONS:
Procedure: Hyperthermic Intraperitoneal Chemotherapy — HIPEC is a way of intraperitoneal chemotherapy
  Arms: Hyperthermic Intraperitoneal chemotherapy

SUMMARY:
This study evaluate the Hyperthermic Intraperitoneal Chemotherapy(HIPEC) in the treatment of Stage IIc-IV epithelial Ovarian Cancer after primary Cytoreductive Surgery (CRS).Half participants will receive HIPEC twice with one intravenous chemotherapy and 5 cycles of intravenous chemotherapy with carboplatin and paclitaxel after CRS. Half participants will receive 6 cycles of intravenous chemotherapy with carboplatin and paclitaxel after CRS.

DETAILED DESCRIPTION:
Advanced epithelial ovarian cancer, now recognized as the most effective treatment is maximizing tumor reduction (cytoreductice surgery, CRS) within the abdominal cavity with platinum-based chemotherapy (intraperitoneal chemotherapy, IPEC) or intravenous chemotherapy.

Hyperthermic intraperitoneal chemotherapy (HIPEC) refers to the chemotherapy drugs will be diluted and heated to the specified temperature (usually the 42 degrees), then injected into the abdominal cavity, maintain a constant temperature, repeated perfusion filling, so as to achieve the purpose of prevention and treatment of intra-abdominal tumors of a way of treatment.

CRS combined with HIPEC is the most effective treatment strategy for peritoneal cancer at present.

ELIGIBILITY:
Inclusion Criteria:

1. the patient voluntarily joined the study and signed the consent form;
2. female patients aged between 18 and 70 who are not pregnant or lactating;
3. primary epithelial ovarian cancer, fallopian tube cancer and primary peritoneal cancer were diagnosed at the time of diagnosis, and no chemotherapy or radiotherapy was given within three months before the study began;
4. laparoscopic Fagotti score <6;
5. residual lesions in abdominal cavity after tumor cell extinction <1cm;
6. expected survival time ≥12 weeks;
7. ECOG score: 0-1;
8. bone marrow reserve function is good, and blood routine indexes meet the following requirements: white blood cell count ≥3.0×109/L, neutrophil absolute count ≥1.5×109/L, platelet count ≥100×109/L, hemoglobin ≥90 g/L;
9. important organs function well and blood biochemical indexes meet the following requirements: serum albumin ≥30 g/L, ALT≤2.5× normal upper limit (ULN), AST≤2.5×ULN, serum total bilirubin ≤1.5×ULN, serum creatinine ≤1.5×ULN.

Exclusion Criteria:

1. refuse to sign the informed consent;
2. other malignant tumors in the past 5 years or at the same time, except cured basal cell carcinoma of skin, cervical carcinoma in situ, thyroid papillary carcinoma and breast cancer without recurrence 3 years after radical resection;
3. laparoscopic Fagotti score ≥6;
4. extensive adhesion exists in the abdominal cavity.
5. >1cm of residual lesions in the abdominal cavity after tumor cell extinction;
6. patients with previous gastrointestinal perforation, abdominal abscess or recent intestinal obstruction (within 3 months), or with imaging and clinical symptoms indicating intestinal obstruction;
7. suffer from other difficult to control serious diseases, including uncontrolled hypertension, NYHA grade 2 or above heart failure, unstable angina, atrial fibrillation, myocardial infarction (within the previous 1 year), renal insufficiency, uncontrollable infection, etc.;
8. significant clinically significant bleeding symptoms and abnormal coagulation function (INR>2.0 or prothrombin time >16s) within the previous 3 months, with a clear tendency to bleeding or being treated with thrombolysis or anticoagulant therapy;
9. occurrence of thrombotic events in the past six months, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism;
10. congenital or acquired immune deficiency;
11. with active hepatitis, active ulcer, unhealed wound or fracture;
12. being treated with other anticancer drugs;
13. the investigator assessed and determined that there were any other unstable conditions, including alcohol abuse, drug abuse, other family or social factors, that might affect patient safety and compliance or cause the study to be discontinued.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the progression-free survival (PFS) of patients with advanced ovarian cancer undergoing primary tumor cell depletion (HIPEC) during surgery. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  From the date of random enrollment to the date of tumor progression or death. The appearance of the new lesion was taken as the criterion of progression, and the date of the first measurable observation of the new lesion was the marker of progression.ovarian cancer undergoing primary tumor cell depletion (HIPEC) during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: JIONG MA, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital, Zhejiang University, School Of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No